## **COVER PAGE**

Title: Acinetobacter baumannii - related osteomyelitis: clinical and epidemiological

characterization

NCT number: NCT03559530

Date: 08/18/2020

**FINAL REPORT** 

Study title: Acinetobacter baumannii - related osteomyelitis: clinical and epidemiological

characterization

**Pfizer Tracking Number: WI176466** 

The initial database consisted of 262 patients with bone tissue culture positive for

Acinetobacter baumannii submitted to surgical procedures to treat osteomyelitis at the Instituto

de Ortopedia e Traumatologia da HCFMUSP from January 2007 to December 2015. From this

total, it was possible to collect data for 171 patients for analysis. Here is a description of the

reason for not including 91 patients:

- non-location of medical records: 44 patients;

- culture results were not considered for treatment: 29 patients;

- duplicate cases in the database: 8 patients;

- cultures showing other species of *Acinetobacter*: 7 patients;

- cultures harvested at the time of initial treatment of cases of exposed fractures and

considered as contamination / colonization: 3 patients.

The descriptive analysis of the total sample (171 patients) and the result of the

comparison between the cases of patients with extensively drug resistant (XDR) isolates treated

with tigecycline and colistin (65 patients) are described in the following report and represents

the largest case series of osteomyelitis related to A. baumannii ever described. The study

protocol was registered in clinicaltrials.gov (NCT03559530).

## 1. Descriptive analysis of the Acinetobacter baumannii osteomyelitis database

- 1.1. Demographics of 171 patients (percentage and absolute numbers)
- Average age: 43.2 years
- Male sex: 78.4% (134)
- Any comorbidity present: 33.9% (58)
  - o Sistemic hypertension: 21.1% (36)
  - Neoplasia: 3.5% (6)
  - o Diabetes mellitus: 10.5% (18)
  - HIV infection: 1.2% (2)
  - o Rheumatoid arthritis: 4.7% (8)
  - Systemic lupus erythematosus: 0.6% (1)
  - Other rheumatological conditions: 1,2% (2)
  - Use of immunosuppressive drugs: 3.5% (6)
- Epidemiological background
  - o Smoking: 6.4% (11)
  - Alcohol abuse: 5.8% (10)
  - Ilicit drug use: 0.6% (1)
  - o Previous surgical site infection in the affected segment: 25.1% (43)
  - o Prior orthopedic surgery: 43.3% (74)
- Affected segment
  - o Hip: 24.6% (42)

- o Leg: 21.6% (37)
- o Thigh: 15.8% (27)
- o Spine: 14.6% (25)
- Foot and ankle: 9.4% (16)
- o Knee: 8.2% (14)
- o Arm: 2.3% (4)
- o Forearm: 1.8% (3)
- Hand and wrist: 1.2% (2)
- o elbow: 0.6% (1)
- Co-infection agents present: 72.5% (124)
  - o S. aureus: 19.4% (24)
  - o Coagulase-negative Staphylococcus spp.: 19.4% (21)
  - o Klebsiella pneumoniae: 16.1% (20)
  - o Pseudomonas aeruginosa: 17.7% (22)
  - o *Candida* spp .: 0.8% (1)
  - o *Enterococcus* spp .: 28.2% (35)

• Antibiogram of A. baumannii isolates for the 171 patients included (table 1).

Table 1 - Antibiogram for A. baumannii samples from the 171 patients included.

| Antimicrobial | Susceptibility | Not tested |
|----------------------|----------------|------------|
| Amikacin | 61,4% (105) | 0,6% (1) |
| Ampicillin/sulbactam | 43,3% (74) | 0% (0) |
| Cefepime | 15,8% (27) | 1,2% (2) |
| Ceftazidime | 14% (24) | 5,8% (10) |
| Ciprofloxacin | 14,6% (25) | 5,8% (10) |
| Imipenem | 35,1% (60) | 0,6% (1) |
| Meropenem | 33,3% (57) | 4,1% (7) |
| Colistin | 63,7% (109) | 33,9% (58) |
| Tigecycline | 47,4% (81) | 38% (65) |
| Gentamicin | 58,5% (100) | 0% (0) |

Table 2 and Figures 1 to 7 below show the evolution of the susceptibility profiles of *A. baumannii* isolates against the main antimicrobials tested during the period in which the patients included in the study were treated. Tigecycline is not included in this analysis because A. baumannii susceptibility to this antimicrobial was extrapolated from breakpoints for enterobacteria during the study period, according to Clinical and Laboratory Standards Institute (CLSI) criteria.

 Table 2 – Percentage of A. baumannii isolates susceptible to main antimicrobials tested during the study period

| | Amikacin | Ampi/Sulb | Cefepime | Ceftazidime | Ciprofloxacin | Carbapenem | Gentamicin |
|---|---|---|---|---|---|---|---|
| 2007 | 29 | 79 | 14 | 14 | 14 | 43 | 50 |
| 2008 | 23 | 73 | 14 | 9 | 9 | 55 | 45 |
| 2009 | 29 | 59 | 18 | 18 | 12 | 47 | 76 |
| 2010 | 79 | 37 | 5 | 11 | 11 | 37 | 53 |
| 2011 | 58 | 27 | 19 | 15 | 15 | 27 | 65 |
| 2012 | 80 | 50 | 25 | 20 | 25 | 45 | 55 |
| 2013 | 84 | 29 | 16 | 16 | 16 | 26 | 68 |
| 2014 | 91 | 18 | 9 | 9 | 9 | 9 | 36 |
| 2015 | 82 | 18 | 18 | 9 | 18 | 18 | 64 |



Figure 1 – Evolution of the susceptibility profile of isolates of A. baumannii to amikacin over study period



**Figure 2** – Evolution of the susceptibility profile of isolates of *A. baumannii* to ampicillin/sulbactan over study period



Figure 3 – Evolution of the susceptibility profile of isolates of A. baumannii to cefepime over study period



Figure 4 – Evolution of the susceptibility profile of isolates of A. baumannii to ceftazidime over study period



Figure 5 – Evolution of the susceptibility profile of isolates of A. baumannii to ciprofloxacin over study period



**Figure 6** – Evolution of the susceptibility profile of isolates of *A. baumannii* to carbapenems (imipenem and meropenem) over study period



Figure 7 – Evolution of the susceptibility profile of isolates of A. baumannii to gentamicin over study period

## • Classification of osteomyelitis

o Post traumatic: 64.9% (111)

o Contiguous: 29.8% (51)

o Spine osteomyelitis: 2.9% (5)

| o Hematogenic: 2.3% (4) |
|---|
| o Acute: 52.6% (90) |
| o Chronic: 47.4% (81) |
| <ul> <li>Previous open fracture: 36.8% (63). Open fracture classification according to Gustilo and</li> </ul> |
| Anderson |
| <ul> <li>No registeredclassification: 22.2% (14)</li> </ul> |
| o II: 4.8% (3) |
| o IIIa: 14.3% (9) |
| o IIIb: 44.4% (28) |
| o IIIc: 14.3% (9) |
| • Neuropathic foot infection: 2.9% (5) |
| • Decubitus ulcer infection: 16.4% (28) |
| • Closed fracture: 9.4% (16) |
| • ASA score: |
| o ASA I: 35.1% (60) |
| o ASA II: 51.5% (88) |
| o ASA III: 13.5% (23) |
| • need for muscle or skin flap repair during osteomyelitis treatment: 32.2% (55) |
| • Negative pressure therapy: 25.1% (43) |
| • Hyperbaric oxygen therapy: 1.2% (2) |

• Average number of surgical procedures for treatment: 3.5

## Antimicrobial use

- o Prior to diagnosis of A. baumannii infection: 90.6% (155)
- o Use of combination therapy (two active drugs) for A. baumannii: 2.9% (5)
- o Treatment groups:
  - o Colistin: 19.9% (34)
  - o Ampicillin / Sulbactam: 18.7% (32)
  - Tigecycline: 18.1% (31)
  - o Aminoglycosides: 15.2% (26)
  - o Quinolone: 14% (24)
  - Carbapenem: 10.5% (18)
  - Aminoglycoside + tigecycline: 1.2% (2)
  - Aminoglycoside + Colistin: 0.6% (1)
  - 3th and 4th generation cephalosporins: 0.6% (1)
  - Sulfamethoxazole / trimethoprim: 0.6% (1)
  - Tigecycline + Colistin: 0.6% (1)
- OPAT: 14% (24)
- Average length of antimicrobial treatment time: 72.6 days
- Average length of hospital stay: 77.9 days
- Adverse events
  - o Some adverse event: 21.6% (37)
  - o Change of microbial drug due to adverse event: 3.5% (6)

• Outcome

After 1 year (favorable X unfavorable)

o Favorable: 53.8% (92)

After 1 year (detailed)

o Remission: 53.8% (92)

Relapse: 15.2% (26)

Amputation: 14.6% (25)

Loss of follow-up: 12.3% (21)

Death related to A. baumannii infection: 3.5% (6)

Death not related to A. baumannii infection: 0.6% (1)

2. Comparative analysis of cases of osteomyelitis by A. baumannii XDR treated with

either colistin or tigecycline

For this analysis, the 65 patients with XDR A. baumannii -related osteomyelitis, always

resistant to carbapenems, treated with colistin or tigecycline were included. The choice of

antimicrobial was at the discretion of the attending physicians responsible for each patient

during their hospitalization and was not influenced by this study, since this is a retrospective

analysis.

Baseline characteristics of each group were compared, according to:

- demographic variables and clinical characteristics already described above,

- tincidence of adverse events related to the treatment and

- outcomes of the patients according to the antimicrobial used.

Quantitative characteristics were described according to groups using summary

measures (mean ± standard deviation or median (minimum; maximum) and compared between

groups using Student's t-tests or Mann-Whitney tests. Qualitative characteristics of the patients

were described according to groups using absolute and relative frequencies, association between groups were tested using chi-square or exact tests (Fisher's exact test or likelihood ratio test). The software used for the analysis was Microsoft-SPSS for Windows version 20.0. Microsoft Excel 2003 was the software used for data tabulation. Tests were performed at a significance level of 5%.

Table 3 shows the distribution of the 65 patients according to each treatment group (colistin or tigecycline) regarding demographic variables and clinical characteristics. In the group of patients treated with tigecycline, the frequency of men was statistically lower than in the group treated with colistin (p = 0.028). In the group of patients treated with tigecycline, there were also predominance of smokers (p = 0.021) and patients with chronic osteomyelitis (p = 0.036).

**Table 3** - Distribution of patients with XDR *A. baumannii* osteomyelitis according to demographic and clinical characteristics and comparison according to treatment group (colistin or tigecycline).

| Mariable | Treati | - Tatal (N - CE) | _ | |
|---|---|---|---|---|
| Variable | Colistin (N = 34) | Tigecycline (N = 31) | Total (N = 65) | р |
| Sex (Male) | 29 (85,3) | 19 (61,3) | 48 (73,8) | 0,028 |
| Age (years) | 40,6 ± 19,1 | 46,8 ± 18,9 | 43,6 ± 19,1 | 0,193** |
| Length of hospital stay (days) | 74,5 (13; 331) | 64 (0; 226) | 70 (0; 331) | 0,948£ |
| Charlson index | 0 (0; 5) | 1 (0; 7) | 0 (0; 7) | 0,083£ |
| Presence of comorbidity | 10 (29,4) | 13 (41,9) | 23 (35,4) | 0,292 |
| Systemic hypertension | 6 (17,6) | 9 (29) | 15 (23,1) | 0,277 |
| Neoplasia | 2 (5,9) | 3 (9,7) | 5 (7,7) | 0,663* |
| Diabetes | 4 (11,8) | 2 (6,5) | 6 (9,2) | 0,674* |
| HIV | 0 (0) | 2 (6,5) | 2 (3,1) | 0,224* |
| Rheumatoid arthritis | 2 (5,9) | 1 (3,2) | 3 (4,6) | >0,999* |
| Systemic lupus erythematosus | 0 (0) | 0 (0) | 0 (0) | а |
| Ankylosing spondylitis | 0 (0) | 0 (0) | 0 (0) | а |
| Other rheumatic diseases | 0 (0) | 1 (3,2) | 1 (1,5) | 0,477* |
| Use of immunosuppressive drugs | 1 (2,9) | 1 (3,2) | 2 (3,1) | >0,999* |
| Chemotherapy | 0 (0) | 0 (0) | 0 (0) | а |
| Chronic Renal Disease | 0 (0) | 0 (0) | 0 (0) | a |
| Previous SSI in the affected segment | 10 (29,4) | 7 (22,6) | 17 (26,2) | 0,531 |
| Injectable drug abuse | 0 (0) | 1 (3,2) | 1 (1,5) | 0,477* |
| Smoking | 0 (0) | 5 (16,1) | 5 (7,7) | 0,021* |
| Alcohol abuse | 2 (5,9) | 4 (12,9) | 6 (9,2) | 0,413* |
| Previous orthopedic surgery in the affected segment | 10 (29,4) | 14 (45,2) | 24 (36,9) | 0,189 |
| Affected Segment | | | | 0,414 |
| Lower limbs | 29 (85,3) | 24 (77,4) | 53 (81,5) | |
| Upper limbs | 5 (14,7) | 7 (22,6) | 12 (18,5) | |
| Other agents detected | 24 (70,6) | 21 (67,7) | 45 (69,2) | 0,804 |

| Classification of osteomyelitis Lima and Zumiotti | | | | 0,841# |
|---|---|---|---|---|
| Post-traumatic | 23 (67,6) | 19 (61,3) | 42 (64,6) | |
| Contiguity | 7 (20,6) | 9 (29) | 16 (24,6) | |
| Hematogenic | 2 (5,9) | 2 (6,5) | 4 (6,2) | |
| Spine | 2 (5,9) | 1 (3,2) | 3 (4,6) | |
| Time classification of osteomyelitis | | | | 0,036 |
| Acute | 22 (64,7) | 12 (38,7) | 34 (52,3) | |
| Chronic | 12 (35,3) | 19 (61,3) | 31 (47,7) | |
| Antecedent of open fracture | 17 (50) | 10 (32,3) | 27 (41,5) | 0,147 |
| Infection in pressure ulcer | 6 (17,6) | 4 (12,9) | 10 (15,4) | 0,736* |
| Antecedent of closed fracture | 1 (2,9) | 4 (12,9) | 5 (7,7) | 0,184* |
| ASA Classification | | | | 0,189 |
| 1 | 11 (32,4) | 8 (25,8) | 19 (29,2) | |
| II | 20 (58,8) | 15 (48,4) | 35 (53,8) | |
| III | 3 (8,8) | 8 (25,8) | 11 (16,9) | |
| Number of surgical procedures for treatment | 3 (1; 12) | 3 (1; 9) | 3 (1; 12) | 0,510£ |
| Presence of implant | 6 (17,6) | 3 (9,7) | 9 (13,8) | 0,480* |
| Need to remove the implant | 4 (11,8) | 9 (29) | 13 (20) | 0,082 |
| Need for soft tissue repair | 10 (29,4) | 8 (25,8) | 18 (27,7) | 0,746 |
| Use of negative pressure therapy | 12 (35,3) | 6 (19,4) | 18 (27,7) | 0,151 |
| Hyperbaric oxygen use | 1 (2,9) | 0 (0) | 1 (1,5) | >0,999* |
| Pain | 6 (17,6) | 7 (22,6) | 13 (20) | 0,619 |
| Hyperemia | 9 (26,5) | 4 (12,9) | 13 (20) | 0,172 |
| Local elevated temperaure | 2 (5,9) | 1 (3,2) | 3 (4,6) | >0,999* |
| Fistula | 19 (55,9) | 19 (61,3) | 38 (58,5) | 0,659 |
| Edema | 1 (2,9) | 4 (12,9) | 5 (7,7) | 0,184* |
| Fever | 4 (11,8) | 9 (29) | 13 (20) | 0,082 |
| Use of antimicrobial before A. baumannii infection | 34 (100) | 30 (96,8) | 64 (98,5) | 0,477* |
| Other antimicrobials used | 29 (85,3) | 23 (74,2) | 52 (80) | 0,264 |
| Need for OPAT | 4 (11,8) | 9 (29) | 13 (20) | 0,082 |
| Baseline Creatinine | $0,69 \pm 0,36$ | $0.82 \pm 0.54$ | 0,75 ± 0,45 | 0,260** |
| Full treatment lenght (days) | 42,5 (1; 193) | 42 (9; 193) | 42 (1; 193) | 0,438£ |

Data expressed as n (%), mean ± SD or median (min, max.); Chi-square test; \* Fisher's exact test; # Likelihood ratio test; \*\* Student's t-test; £ Mann-Whitney test; a There are no cases to estimate

Regarding the registered adverse events, table 4 shows the comparison between the two treatment groups. It is possible to observe that the general incidence of adverse events was higher in the group of patients treated with colistin (p = 0.047), as well as the incidence of renal impairment (p = 0.003). The incidence of nausea and vomiting was higher in the group of patients treated with tigecycline (p = 0.046).

Table 4 - Comparison of incidence of adverse events during treatment for patients receiving colistin or tigecycline

| Variable | Treatr | Total (N = 65) | р | |
|---|---|---|---|---|
| | Colistin (N = 34) | Colistin (N = 34) Tigecycline (N = 31) | | |
| Overall adverse events | 23 (67,6) | 13 (41,9) | 36 (55,3) | 0,047 |
| Renal impairment | 20 (58,8) | 7 (22,6) | 27 (41,5) | 0,003 |
| Liver abnormalities | 1 (2,9) | 1 (3,2) | 2 (3,1) | >0,999* |
| Nausea | 0 (0) | 4 (12,9) | 4 (6,2) | 0,046* |
| Neural alterations | 0 (0) | 0 (0) | 0 (0) | a |
| Skin rash | 1 (2,9) | 0 (0) | 1 (1,5) | >0,999* |
| Other | 5 (14,7) | 2 (6,4) | 7 (10,7) | 0,430 |

Data expressed as n (%) or mean ± SD; Chi-square test; \* Fisher's exact test; \*\* Student's t-test; a There are no cases to estimate

Due to the characteristics of the osteomyelitis evolution, the treatment outcome was assessed based on the patient's evaluation 12 months after the end of the treatment. Evaluated outcomes were remission of the infection (absence of signs and symptoms compatible with osteomyelitis activity), relapse (patient returning with signs and symptoms of infection up to 12 months after treatment), amputation, death and loss of follow-up. The outcomes were also evaluated in a dichotomous way, being considered remission as a favorable outcome and recurrence, amputation and death and as unfavorable outcomes. Patients who presented loss of follow-up were analyzed in two ways: as a separate outcome and as part of unfavorable outcomes. There were no significant differences between the two treatment groups in these analyzes, as can be seen in Tables 5 and 6.

Table 5 - Distribution of the outcomes after 12 months of treatment according to the antimicrobial group

| Outcome | Treatn | Total (N = 65) | <b>n</b> | |
|---|---|---|---|---|
| | Colistin (N = 34) | Tigecycline (N = 31) | 10tai (N - 65) | р |
| Remission | 15 (44,1) | 12 (38,7) | 27 (41,5) | 0,801 |
| Death | 2 (5,8) | 3 (9,6) | 5 (7,7) | 0,663 |
| Recidive | 5 (14,7) | 6 (19,3) | 11 (16,9) | 0,744 |
| Amputation | 7 (20,6) | 2 (6,45) | 9 (13,8) | 0,152 |
| Loss of follow-up | 5 (14,7) | 8 (25,8) | 13 (20) | 0,355 |

Data expressed as n (%); Chi-square test to estimate

**Table 6** - Dichotomic distribution of the outcomes after 12 months of treatment according to the antimicrobial group

| Outcome | Treatr | nent group | T-1-1/N CF) | |
|---|---|---|---|---|
| | Colistin (N = 34) Tigecycline (N = 31) | | Total (N = 65) | р |
| Outcome | | - | _ | 0,535 |
| Unfavorable | 14 (41,2) | 11 (35,5) | 25 (38,5) | |
| Favorable | 15 (44,1) | 12 (38,7) | 27 (41,5) | |
| Loss of follow-up | 5 (14,7) | 8 (25,8) | 13 (20) | |
| Outcome | | | | 0,659 |
| Unfavorable | 19 (55,9) | 19 (61,3) | 38 (58,5) | |
| Favorable | 15 (44,1) | 12 (38,7) | 27 (41,5) | |

Data expressed as n (%); Chi-square test to estimate

Analysis of presented data allows us to conclude that, in this sample of patients studied, tigecycline presented a better safety profile than colistin for the treatment of osteomyelitis related to XDR carbapenem resistant *A. baumannii*. Both antimicrobial presented similar efficacy. The data presented in this report will be submitted for scientific publication.